CLINICAL TRIAL: NCT07139990
Title: Personalized Radiotherapy for Individualized Treatment Strategies and Monitoring (PRISM): A Multi-cohort Platform Trial of Adaptive Radiotherapy Approaches in Multiple Cancer Types
Brief Title: Personalized Radiotherapy for Individualized Treatment Strategies and Monitoring (PRISM)
Acronym: PRISM
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Neil Desai, Principal Investigator, MD MHS, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20251050
Record Dates: First submitted 2025-08-12; First posted 2025-08-24 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Small Cell Lung Cancer Extensive Stage; Brain Metastases; Solid Tumor, Adult
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: Cohort A: >= 18 yo with extensive stage small cell lung cancer receiving standard chemoimmunotherapy and eligible for thoracic radiotherapy Cohort B: >= 18 yo with solid tumor brain metastases (<=5 total; size>=2cm in brain or >=1.5cm in brainstem) planned for fractionated stereotactic radiotherapy (fSRT)
Masking Description: n/a No radiotherapy will be given aside from standard of care. However, this study will focus on compressing the time frame in which said therapy is administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COHORT A (ES-SCLC PULSAR Thoracic Tumor): (Experimental): PULSAR with online adaptive planning to 7-10 Gy per fraction for up to 3 pulses directed at the bulkiest sites of disease in the thorax before infusion days (window: D-1 to D-4; optimal D-1) of three cycles of chemoimmunotherapy. The first radiotherapy pulse must be delivered before chemoimmunotherapy cycle 4. The three "pulses" of radiotherapy ideally should be given with consecutive cycles of systemic therapy. Radiotherapy can be suspended if a complete clinical response is reached before all 3 pulses are delivered. Chemoimmunotherapy will be given per standard of care
  Interventions: Radiation: Cohort A: Extensive Stage Small Cell Lung Cancer (ES-SCLC) Thoracic Tumor PULSAR (Personalized ultrahypofractionated stereotactic ablative radiotherapy)
- COHORT B (Brain metastasis PULSAR): (Experimental): PULSAR will be delivered in a 2 "pulse" strategy:
  1: Deliver fSRT/SRS every other day (minimum 48 hour separation between treatments, minimum 1 treatment per week;begin and complete within 60 days of registration) for 3 fractions. Pulse 1 must begin and complete within 60 days of registration; 2) Repeat treatment planning MRI will be performed after 4 weeks (window: +/-1 weeks) after fraction 3 and volumetric response assessment made; 3) Pulse 2 is omitted in those with >=25% volumetric size reduction response. In others, pulse 2 will deliver fSRT/SRS every other day (minimum 48 hour separation between treatments, minimum 1 treatment per week). Pulse 2 may deliver higher dose per fraction within Section 4.1.3.4 specifications (Table 6), rationale for this would be for addressing lesions that either due to large size or proximity to critical structures could only be treated to a lower dose range in pulse 1. Pulse 2 must begin 4 weeks (+/-1 weeks) after end of Pulse 1.
  Interventions: Radiation: Cohort B: Brain metastasis PULSAR (Personalized ultrahypofractionated stereotactic ablative radiotherapy)

INTERVENTIONS:
Radiation: Cohort A: Extensive Stage Small Cell Lung Cancer (ES-SCLC) Thoracic Tumor PULSAR (Personalized ultrahypofractionated stereotactic ablative radiotherapy) — Radiographic response-adapted thoracic tumor radiotherapy given as single doses ('pulses') before standard of care chemoimmunotherapy cycles. Adaptive Changes Allowed: Tumor target (size/shape), # of doses (reduction) Adaptive Changes Allowed: Tumor target (size/shape), # of doses (reduction)
  Arms: COHORT A (ES-SCLC PULSAR Thoracic Tumor):
Radiation: Cohort B: Brain metastasis PULSAR (Personalized ultrahypofractionated stereotactic ablative radiotherapy) — Intervention: Fractionated stereotactic radiosurgery (SRS, 5 doses total) for brain metastasis given in two "pulses" (3 fractions + 2 fractions) with second pulse adapted to interim radiographic response Adaptive Changes Allowed: Omission of 2nd "pulse" in >=25% responders or tumor target size/shape change in remainder
  Arms: COHORT B (Brain metastasis PULSAR):

SUMMARY:
To characterize feasibility, safety, and/or preliminary efficacy of personalized strategies to adapt standard radiotherapy treatments to individual patient responses.

DETAILED DESCRIPTION:
Cohort-Specific Rationale

COHORT A (ES-SCLC Personalized ultrahypofractionated stereotactic ablative radiotherapy (PULSAR) Thoracic Tumor):

Chemoimmunotherapy with 4-6 cycles of platinum/etoposide and PD-L1 (Programmed Death-Ligand 1 protein) inhibition has become the standard systemic therapy for extensive stage small cell lung cancer (ES-SCLC), based on modest but significant OS (overall survival) benefits seen with the addition of either atezolizumab or durvalumab to chemotherapy in the IMpower133 and CASPIAN trials, respectively. However, outcomes remain poor with median OS of only 12.3 months. Notably, consolidative thoracic RT (radiotherapy) was not allowed either trial. This contrasts with prior signal for potential benefit for addition of thoracic RT to standard chemotherapy in ES-SCLC in the CREST trial, though this was not duplicated the RTOG 0937. Encouraging preliminary safety data has been published for addition of hypofractionated thoracic RT to single agent PD-1 inhibition after response to induction chemotherapy (6% grade 3 toxicity), but toxicities with doublet immune checkpoint blockade (ipilimumab/nivolumab) and RT showed a nearly 20% rate of high grade AEs (adverse events). This has led to an ongoing cooperative study (NRG LU007) seeking to define the impact of consolidative thoracic RT given with atezolizumab following induction chemotherapy. In the interim, while use of thoracic RT consolidation in ES-SCLC remains supported as a standard of care by guidelines, its implementation is variable. Particularly important open question involve timing for synergy/additivity with immune checkpoint blockade and cytotoxic therapy, minimization of target size for safety, and tailoring of dose according to patient need given significant competing risks for extra-thoracic progression and tolerance. In seeking to address this, this study notes that small cell lung cancer generally shrinks rapidly with each cycle of chemoimmunotherapy. Delivering a "pulse" of RT to the thoracic disease immediately prior to cycles 2-6 of chemoimmunotherapy may result in faster tumor response and reduction of overall treatment target size. Moreover, prolongation of time between doses enables observation of response, which would allow investigators to withhold further RT dose in those unlikely to benefit due to extra-thoracic progression or exceptional early response of thoracic disease.

COHORT B (Brain metastasis PULSAR):

Brain metastases from solid tumors affect nearly 30% of patients who die of cancer and present an increasing challenge for management as patients live longer with improved systemic therapies. Treatment often includes radiotherapy, increasingly delivered as stereotactic radiosurgery (SRS) to spare normal brain. For larger lesions or those near sensitive areas, fractionated stereotactic radiation therapy (FSRT) delivered in up to 5 treatments is used to reduce swelling and late injury. Prolongation of the duration between fSRT treatments from days to weeks further has enabled adjustments of the treatment target to tumor size changes over treatment, further reducing healthy brain exposure without sacrifice in tumor control (7). UT Southwestern has expanded upon this modified fSRT approach with PULSAR. Based upon observed kinetics of response, the predominant PULSAR approach has been to deliver treatments in two "pulses" given as 3 fractions every other day, 3-4 week break, and then 2 final fractions every other day. In the initial experience (n=109 treated lesions), PULSAR demonstrated favorable efficacy and tolerability in treating brain metastases (2-year 90% local control and <10% grade 3 toxicity), when compared to historical fSRT reports especially for larger >=2cm lesions. PULSAR for brain metastases thus shows high potential to address larger tumors and to individualize RT dose/intensity, especially in the setting of increasing numbers of central nervous system (CNS)-active systemic agents.

In particular, with longer patient survivals, there remains a critical need to reduce the risk of toxicity and edema by de-escalating dose in addition to target size. The best 'biomarker' for such de-escalation appears to be early radiographic response, with published work strongly correlating a >=20% lesion volume reduction by 3-months to improved local control. Notably, such reductions are commonly seen in time for decision making in the PULSAR approach, with the collected data previously showing a median 38% reduction in larger tumors (>=2cm) during treatment. Specifically, ~50% of patients achieve a 25% reduction by pulse 2. In this cohort, the study will assess whether a more conservative >=25% tumor volume at interim imaging of PULSAR can be used to omit the second "pulse" for "responders," while retaining high control rates.

ELIGIBILITY:
Inclusion Criteria:

Cohort A:

* >=18 years old
* Performance status ECOG 0-2
* Extensive stage small cell lung cancer diagnosed by tissue biopsy within 180 days of registration.
* Patient must be planned for or receiving standard of care chemoimmunotherapy.
* Patient must have received no more than 3 cycles by time of study enrollment.
* Able and indicated according to investigator to receive thoracic radiotherapy

Cohort B:

* 18 years old
* Diagnosis of solid tumor malignancy with MRI-defined brain metastasis lesions (1-5 lesions allowed) within 60 days of registration
* Each brain metastasis lesion enrolled must be 2 - 5 cm, except brainstem lesions which may be 1.5 - 5cm in size.

Exclusion Criteria:

Cohort A:

⨀ Prior thoracic Radiotherapy

Cohort B:

* Prior whole brain Radiotherapy
* Prior surgical resection or focal radiotherapy of a target brain metastasis
* Leptomeningeal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
COHORT A-assess safety of addition of PULSAR radiotherapy to thoracic tumor in ES-SCLC alongside chemoimmunotherapy, while making preliminary/exploratory assessments of disease response and dosimetric benefit to PULSAR | 5 years
  Primary objective will be to report safety of PULSAR with chemoimmunotherapy for extensive stage small cell lung cancer. Accrual goal will be 15 patients.Study is interested in precise estimates of safety as well as outcome variability that will aid in the planning of larger, sufficiently powered efficacy trial. Sample size of 15 patients will allow for relative precision in conclusions regarding safety outcome.Namely,if 4 out of 15 patients enrolled are observed as having grade 3+ cardiopulmonary acute toxicity,the 95% CI for that rate would be (7.95%-55.10%) using an Exact (Clopper-Pearson) binomial confidence interval.
  Descriptive statistics according to variable type (continuous, categorical) will be used for reporting the cohort characteristics. Primary endpoint of pre-defined high grade toxicities will be reported as a categorical percentage.Disease control(time to event variables) will be reported by Kaplan-Meier estimates.
COHORT B-assesses ability to de-escalate dose in good responders by imaging using rule-based imaging-response guided omission of 2nd "pulse" of PULSAR fractionated SRS (fSRS) for brain metastases | 5 years
  Sample size comparing local control & toxicity with prior PULSAR data(which didn't dose de-escalate based on response)to ensure high control rate is preserved.Using two-tailed test with alpha of 0.05 & power of 0.8,estimated sample size to detect difference in 1-yr local failure rates between pSRT & fSRT.Stats according to variable type(continuous,categorical)used for reporting primary endpoint of proportion of patients de-escalated & endpoints.To evaluate local control & toxicity(late CNS),competing risk regression & calculated cumulative incidence,with death as competing risk will be performed.Gray's test will be used to assess statistical significance.OS analyzed using Kaplan-Meier method using survival,log-rank test employed to compare survival distributions.To account for clustered data,where patients may have multiple brain metastases treated,repeated analyses for CRR using crrSC(R package)will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: NEIL DESAI, MD, MHS, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Ut Southwestern Medical Center, Dallas, Texas, United States